CLINICAL TRIAL: NCT06455618
Title: The Feasibility, Safety, and Efficacy of Not Indwelling of Ureteral Stents in Percutaneous Nephrolithotomy: A Randomized Controlled Trial
Brief Title: The Feasibility, Safety, and Efficacy of Not Indwelling of Ureteral Stents in Percutaneous Nephrolithotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Guohua Zeng, Vice president, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MRER(42)2023
Record Dates: First submitted 2024-06-07; First posted 2024-06-12 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Urolithiasis
Keywords: PCNL; ureteral stent; nephrostomy tube; tubeless; WISQOL questionnaire scores
MeSH Terms: conditions — Urolithiasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- stent-less PCNL (Experimental): In group 1, a nephrostomy tube is indwelled in the patient's body before the end of PCNL.
  Interventions: Procedure: not Indwelling the ureteral stent
- stent PCNL (Active Comparator): In group 2, a nephrostomy tube and a ureteral stent are indwelled in the patient's body before the end of PCNL.
  Interventions: Procedure: Indwelling the ureteral stent

INTERVENTIONS:
Procedure: not Indwelling the ureteral stent — Before the end of surgery, the urologist does not Indwell the ureteral stent in the patient's body. The ureteral stent is usually called "Double-J Stent".
  Arms: stent-less PCNL
Procedure: Indwelling the ureteral stent — Before the end of surgery, the urologist Indwell the ureteral stent in the patient's body. The ureteral stent is usually called "Double-J Stent".
  Arms: stent PCNL

SUMMARY:
Percutaneous nephrolithotomy (PCNL) is currently the preferred treatment for upper urinary tract stones larger than 2cm. In the standard PCNL procedure, a nephrostomy tube and a ureteral stent are often placed before the end of surgery. Recently, PCNL without indwelling nephrostomy tube but with indwelling ureteral stent (also called "tubeless PCNL") or PCNL without indwelling nephrostomy tube and ureteral stent (also called "totally tubeless PCNL") has been put into practice. Compared with the standard PCNL , tubeless or totally tubeless PCNL can effectively reduce postoperative pain and shorten hospital stay, while the incidence of complications does not significantly increase.

Is it possible not to leave a ureteral stent but leave a nephrostomy tube (also called "stent-less PCNL") after PCNL? In theory, the nephrostomy tube can have certain effect, such as decreasing the risk of post-operative bleeding. On the other hand, not indwelling a ureteral stent can bring benefits to patients. Recently, there is limited research on not indwelling ureteral stent after PCNL, and its safety and feasibility require clinical validation.

In summary, investigators conducted a prospective randomized controlled trial to explore the safety and feasibility of not indwelling ureteral stent after PCNL.

DETAILED DESCRIPTION:
Percutaneous nephrolithotomy (PCNL) is currently the preferred treatment for upper urinary tract stones larger than 2cm. In the standard PCNL procedure, a nephrostomy tube and a ureteral stent are often placed before the end of surgery to ensure urine drainage, promote fistula healing, and reduce the occurrence of kidney stones entering the ureter. With the improvement of surgical techniques, PCNL without indwelling nephrostomy tube but with indwelling ureteral stent (also called "tubeless PCNL") or PCNL without indwelling nephrostomy tube and ureteral stent (also called "totally tubeless PCNL") has been put into practice. Compared with the standard PCNL , tubeless or totally tubeless PCNL can effectively reduce postoperative pain and shorten hospital stay, while the incidence of complications does not significantly increase.

Is it possible not to leave a ureteral stent but leave a nephrostomy tube (also called "stent-less PCNL") after PCNL? This clever method combined two advantages. In theory, the nephrostomy tube can have certain effect, such as decreasing the risk of post-operative bleeding, and avoiding the occurrence of emergency events related to ureteral stones. On the other hand, not indwelling a ureteral stent can bring benefits to patients. Recently, there is limited research on not indwelling ureteral stent after PCNL, and its safety and feasibility require clinical validation.

On the other hand, the Wisconsin Stone Quality of Life (WISQOL), as a specific quality of life scoring system for stone patients, has been widely promoted and applied in many countries around the world. Investigators have recently translated this foreign version of the scoring system into Chinese in order to help serve patients with urinary tract stones in China.

In summary, investigators conducted a single center prospective randomized controlled trial (RCT) to compare and analyze the complications of not indwelling ureteral stent after PCNL, WISQOL questionnaire scores, and explore the safety and feasibility of not indwelling ureteral stent after PCNL.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years old
* Renal stones>2cm, preparing for PCNL
* Normal reading comprehension ability

Exclusion Criteria:

* Patients with preoperative neurogenic bladder, Over Active Bladder (OAB), and lower urinary tract symptoms (LUTS).
* Kidney transplantation, isolated kidney, horseshoe kidney, urinary diversion, urinary tract abnormalities.
* Stricture of ureter or stones of the affected ureter require treatment
* Kidney abscess or uncontrolled urinary tract infection
* Internal stent was left in the affected ureter within one year

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-04-02 (Actual); Primary Completion 2024-05-05 (Actual); Study Completion 2024-06-06 (Actual)

PRIMARY OUTCOMES:
Operative time | During surgery
  Surgery duration, minutes
Hospital stay | 1 week
  Duration of hospital stay after surgery, days
Complication rate | 1 month after sugery
  Complication is defined as any adverse event occurred intraoperatively or ≤1 month postoperatively, including intraoperative bleeding, postoperative pain and so on.The investigator will invaluate perioperative complications by modified Clavien system
Visual Analogue Scale(VAS) | 1 day after sugery
  The basic method is to use a moving ruler about 10cm long, with 10 scales on one side and "0" and "10" points on both ends, where 0 represents no pain and 10 represents the most unbearable pain.
Wisconsin Stone Quality of Life questionnaire (WISQOL) Scores | on the 3rd, 14th, and 1st day after surgery
  A total of 28 questions were included in 4 aspects (social, disease, vitality, and emotion), and a questionnaire was recorded and filled out on the 3rd, 14th, and 1st day after surgery through telephone inquiry and evaluation.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Urology, Minimally Invasive Surgery Center, The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China